CLINICAL TRIAL: NCT06315049
Title: Music Therapy to Reduce Anxiety in Community-Dwelling Individuals With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Politècnica de València (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Josep Francesc Silva Galiana, PhD., Universitat Politècnica de València
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-ENFPOD-2621979
Record Dates: First submitted 2024-01-05; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Severe Mental Disorder; Schizophrenia; Bipolar Disorder; Anxiety
Keywords: Music therapy
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music therapy group (Experimental): It is formed from all the participants in the study. They participated in the music therapy sessions.
  Interventions: Other: Music therapy

INTERVENTIONS:
Other: Music therapy — Music therapy sessions to reduce anxiety

SUMMARY:
This study aims to measure the effectiveness of the Music Therapy nursing intervention in reducing anxiety in outpatients diagnosed with severe mental illness (SMI) (bipolar disorder and schizophrenia). The intervention was structured over five weeks (ten 1-hour sessions, twice weekly). Objective measures (blood pressure, heart rate, and respiratory rate) and subjective measures (anxiety response and the subjective perception of relaxation) were taken before and after every session.

DETAILED DESCRIPTION:
This study aims to measure the effectiveness of the Music Therapy nursing intervention in reducing anxiety in outpatients diagnosed with SMI (bipolar disorder and schizophrenia).

The general objective is to evaluate the effectiveness of the Nursing Interventions Classification (NIC) activity, known as Music Therapy, as a therapeutic modality complementary to psychopharmacological treatment for reducing anxiety in patients diagnosed with SMI. The specific research questions are:

Q1: How much do music interventions affect the objective values of vital signs (systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate (HR), and respiratory rate (RR)) in people diagnosed with SMI? Q2: How much does the subjective perception of anxiety change after a music intervention with people diagnosed with SMI? This pilot study is quasi-experimental analytical research of type cross-sectional. It was conducted with outpatients diagnosed with SMI. All patients were recruited from a community mental health center in Valencia (Spain). Fourteen patients regularly attended an occupational activities rehabilitation workshop. All of them were recruited: after the workshop, they participated in the music therapy sessions. All the participants had been previously diagnosed with SMI (schizophrenia, bipolar disorder) by their psychiatrist. Ten participants lived with their parents, and four lived alone and lacked familiar support. None of the participants worked. All had total permanent disability, legally granted, and therefore could not carry out any work activity.

All patients who met the inclusion/exclusion criteria and voluntarily accepted to participate were recruited: 14 patients (3 people with bipolar disorder, 11 people with schizophrenia) participated in the study (with a total sample of 10 group sessions and 150 individual data collection interviews). None of the patients had any previous music therapy experience. All patients followed unique treatments, and this study was an opportunity to motivate their social interaction through music and to study its impact on anxiety.

The patients' psychiatrists determined the cognitive competency of the patients and decided the convenience of their participation.

The intervention was organized into ten 1-hour music therapy sessions at the outpatient level twice weekly. Patients' adherence to the music therapy sessions was 75%, which was more or less stable (standard deviation 15%).

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with SMI (schizophrenia, bipolar disorder) according to the Diagnostic and Statistical Manual of Mental Disorders DSM-V-TR
* currently in outpatient psychiatric treatment in their corresponding mental health unit
* acceptance to enter the study (informed consent); if legally incapacitated, authorization from the patient's legal guardian
* ability to understand the questions in anxiety questionnaires
* between 35 and 50 years of age, to focus the study on a specific population (young adulthood above 35 years and middle adulthood) and to narrow the age range so that they can share common recall of musical memories

Exclusion Criteria:

* suffering from a dual pathology (diagnosis of mental illness and, at the same time, substance abuse) and who were also in the dependency phase
* affected by some type of degenerative disease (dementia, Alzheimer's, etc.)
* presence of positive psychotic symptoms or behavioral disorganization susceptible to admission in the mental health unit
* deafness

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
IDARE test | 1 year
  Inventario de la ansiedad rasgo-estado (IDARE) is the Spanish version of the State-Trait Anxiety Inventory (STAI), commonly used to obtain a meaningful measure of state anxiety (SA) and trait anxiety (TA).
SBP | 1 year
  Systolic blood pressure
DBP | 1 year
  Diastolic blood pressure
HR | 1 year
  Heart rate
RR | 1 year
  Respiratory rate

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Ibáñez, PhD, Study Director — Universitat de València
Locations (1):
- Universitat Politècnica de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibanez-Del Valle V, Sanchez-Martinez V, Silva J. Nurse-Implemented Music Therapy to Reduce Anxiety in Community-Dwelling Individuals with Severe Mental Illness: A Pilot Study. Nurs Rep. 2024 Mar 22;14(2):695-706. doi: 10.3390/nursrep14020053. PMID 38525699